CLINICAL TRIAL: NCT05857943
Title: Prospective Clinical Trial to Demonstrate the Efficacy and Safety if AEYE-DS Software Device for Automated Detection of Diabetic Retinopathy From Digital Funduscopic Images Obtained With a Funduscopic Device
Brief Title: Efficacy and Safety of AEYE-DS Software Device for Automated Detection of Diabetic Retinopathy From Digital Funduscopic Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AEYE Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AEYE-DS-002
Record Dates: First submitted 2023-03-29; First posted 2023-05-15 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AEYE-DS Software Device (Experimental): An AI software device (AEYE-DS) to be used as a diagnostic tool to assist primary care clinicians in screening for diabetic retinopathy using digital funduscopic images. The device automatically detects more than mild diabetic retinopathy (mtmDR) in adults diagnosed with diabetes who have not been previously diagnosed with diabetic retinopathy
  Interventions: Device: AEYE-DS Software

INTERVENTIONS:
Device: AEYE-DS Software — Eligible participants will undergo the following procedures: Photographic imaging of each eye using a funduscopy camera device. Images obtained will be sent to the AEYE-DS software for analysis. -Additional photographic and OCT images will be obtained using a second funduscopy/OCT camera device. Images obtained will be sent to a professional reading center for analysis. -All study subjects will have their pupils dilated using dilation drops.

SUMMARY:
AEYE-DS is a software device developed to increase compliance with diabetic retinopathy screening by automatically detecting more-than-mild diabetic retinopathy from digital funduscopic images using AI-based software. This study has been designed to validate the safety and efficacy of the device at primary care and other point of care sites.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22
2. Male or female
3. Documented diagnosis of diabetes mellitus, meeting the criteria established by the American Diabetes Association (ADA) and World Health Organization (WHO):
4. Understand the study and volunteer to sign the informed consent

Exclusion Criteria:

1. Uncorrectable vision loss (e.g., with the use of eyeglasses), blurred vision, or floaters.
2. Diagnosed with macular edema, severe non-proliferative retinopathy, proliferative retinopathy, radiation retinopathy, or retinal vein occlusion.
3. Previously diagnosed with Diabetic Retinopathy.
4. History of laser treatment of the retina or injections into either eye, or any history of retinal surgery.
5. Currently participating in another investigational eye study and actively receiving investigational product for DR or DME.
6. Participant has a condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure or glycemic control, microphthalmia or previous enucleation).
7. Participant is contraindicated for imaging by fundus imaging systems used in the study:

   1. Participant is hypersensitive to light
   2. Participant recently underwent photodynamic therapy (PDT)
   3. Participant is taking medication that causes photosensitivity
   4. Participant has a history of angle-closure glaucoma or narrow anterior chamber angles
8. Subject is pregnant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Karas Health Care, Fayetteville, Arkansas
  - Lake Nona Research, Orlando, Florida
  - The Jackson Clinic, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: No